CLINICAL TRIAL: NCT03745326
Title: A Phase I/II Study Administering Peripheral Blood Lymphocytes Transduced With a Murine T-Cell Receptor Recognizing the G12D Variant of Mutated RAS in HLA-A*11:01 Patients
Brief Title: Administering Peripheral Blood Lymphocytes Transduced With a Murine T-Cell Receptor Recognizing the G12D Variant of Mutated RAS in HLA-A*11:01 Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 190017; 19-C-0017
Record Dates: First submitted 2018-11-16; First posted 2018-11-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09-22

CONDITIONS: Gastrointestinal Cancer; Pancreatic Cancer; Gastric Cancer; Colon Cancer; Rectal Cancer
Keywords: Immunotherapy; Cell Therapy; KRAS; HRAS; NRAS
MeSH Terms: conditions — Gastrointestinal Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Cyclophosphamide; fludarabine; aldesleukin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Phase I (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + escalating doses of anti-KRAS G12D mTCR PBL + highdose aldesleukin
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Aldesleukin; Biological: anti-KRAS G12D mTCR PBL
- 2/Phase II (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + MTD of anti-KRAS G12D mTCR PBL + high-dose aldesleukin
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Aldesleukin; Biological: anti-KRAS G12D mTCR PBL

INTERVENTIONS:
Drug: Cyclophosphamide — Days -7 and -6: Cyclophosphamide 60 mg/kg/day x 2 days IV in 250 mL D5W infused simultaneously with mesna 15 mg/kg/day over 1 hour x 2 days.
Drug: Fludarabine — Days -7 to -3: Fludarabine 25 mg/m^2/day IVPB daily over 30 minutes for 5 days.
Drug: Aldesleukin — Aldesleukin 720,000 IU/kg IV (based on total body weight) over 15 minutes approximately every 8 hours beginning within 24 hours of cell infusion and continuing for up to 3 days (maximum 9 doses).
Biological: anti-KRAS G12D mTCR PBL — Day 0: Cells will be infused intravenously on the Patient Care Unit over 20-30 minutes (2-4 days after the last dose of fludarabine).

SUMMARY:
Background:

A new cancer therapy takes white blood cells from a person, grows them in a lab, genetically changes them, then gives them back to the person. Researchers think this may help attack tumors in people with certain cancers. It is called gene transfer using anti-KRAS G12D mTCR cells.

Objective:

To see if anti-KRAS G12D mTCR cells are safe and cause tumors to shrink.

Eligibility:

Adults ages 18-72 who have cancer with a molecule on the tumors that can be recognized by the study cells

Design:

Participants will be screened with medical history, physical exam, scans, photography, and heart, lung, and lab tests.

An intravenous (IV) catheter will be placed in a large vein in the chest.

Participants will have leukapheresis. Blood will be removed through a needle in an arm. A machine will divide the blood and collect white blood cells. The rest of the blood will be returned to the participant through a needle in the other arm.

A few weeks later, participants will have a hospital stay. They will:

* Get 2 chemotherapy medicines by IV over 5 days.
* Get the changed cells through the catheter. Get up to 9 doses of a medicine to help the cells. They may get a shot to stimulate blood cells.
* Recover in the hospital for up to 3 weeks. They will provide blood samples.

Participants will take an antibiotic for at least 6 months.

Participants will have several follow-up visits over 2 years. They will repeat most of the screening tests and may have leukapheresis.

Participants blood will be collected for several years.

DETAILED DESCRIPTION:
Background:

* We generated an HLA-A11:01-restricted murine T-cell receptor (mTCR) that specifically recognizes the G12D-mutated variant of KRAS (and other RAS family genes), expressed by many human cancers and constructed a single retroviral vector that contains alpha and beta chains that confer recognition of this antigen when transduced into PBL.
* In co-cultures with HLA-A11:01+ target cells expressing this mutated oncogene, mTCR transduced T-cells lyse target cells and secrete IFN-gamma with high specificity.

Objectives:

-Primary objectives:

* Phase I: Determine the safety of administering PBL transduced with anti-KRAS G12D mTCR in concert with preparative lymphodepletion and high-dose interleukin-2 (IL-2; aldesleukin).
* Phase II: Determine if anti-KRAS G12D mTCR-transduced PBL can mediate the regression of tumors harboring the RAS G12D mutation.

Eligibility:

* Patients must be/have:

  * Age greater than or equal to 18 years and less than or eqaul to 72 years
  * HLA-A*11:01 positive
  * Metastatic or unresectable RAS G12D-expressing cancer which has progressed after standard therapy (if available).
* Patients may not have:

  * Allergies or hypersensitivities to high-dose aldesleukin, cyclophosphamide, or fludarabine.

Design:

* This is a phase I/II, single center study of PBL transduced with anti-KRAS G12D mTCR in HLA-A*11:01 positive patients with advanced solid tumors expressing G12D mutated RAS.
* PBMC obtained by leukapheresis will be cultured in the presence of anti-CD3 (OKT3) and aldesleukin in order to stimulate T-cell growth.
* Transduction is initiated by exposure of these cells to retroviral vector supernatant containing replication-incompetent virus encoding the anti-KRAS G12D mTCR.
* All patients will receive a non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine.
* On Day 0, patients will receive their PBL transduced with the anti-KRAS G12D mTCR and will then begin high-dose aldesleukin.
* A complete evaluation of lesions will be conducted approximately 6 weeks (plus-minus 2 weeks) after treatment.
* The study will be conducted using a phase I/II Simon minimax design, with two separate cohorts for the Phase II component: Cohort 2a, patients with RAS G12D pancreatic cancer, and Cohort 2b, patients with RAS G12D non-pancreatic cancer.
* A total of up to 70 patients may be required; approximately 24 patients in the Phase I portion of the study and 46 (21, plus an allowance of up to 2 non-evaluable per Phase II cohort) patients in the Phase II portion of the study.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Measurable (per RECIST v1.1 criteria), metastatic, or unresectable malignancy expressing G12D mutated KRAS as assessed by one of the following methods: RT-PCR on tumor tissue, tumor DNA sequencing, or any other CLIA-certified laboratory test on

   resected tissue. Patients shown to have tumors expressing G12D mutated NRAS and HRAS will also be eligible as these oncogenes share complete amino acid homology with G12D mutated KRAS for their first 80 N-terminal amino acids, completely encompassing the target epitope.
2. Patients must be HLA-A*11:01 positive as confirmed by the NIH Department of Transfusion Medicine.
3. Confirmation of the diagnosis of cancer by the NCI Laboratory of Pathology.
4. Patients must have:

   -previously received standard systemic therapy for their advanced cancer and have been either non-responders or have recurred, specifically:
   * Patients with metastatic colorectal cancer must have had at least two systemic chemotherapy regimens that include 5FU, leucovorin, bevacizumab, oxaliplatin, and irinotecan (or similar agents), or have contraindications to receiving those medications.
   * Patients with pancreatic cancer must have received gemcitabine, 5FU, and oxaliplatin (or similar agents), or have contraindications to receiving those medications.
   * Patients with non-small cell lung cancer (NSCLC) must have had appropriate targeted therapy as indicated by abnormalities in ALK, EGFR, or expression of PDL-1. Other patients must have had platinum-based chemotherapy.
   * Patients with ovarian cancer or prostate cancer must have had approved first-line chemotherapy.

   OR

   -declined standard treatment.
5. Patients with 3 or fewer brain metastases that are < 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for one month after treatment for the patient to be eligible. Patients with

   surgically resected brain metastases are eligible.
6. Age greater than or equal to 18 years and less than or equal to 72 years.
7. Clinical performance status of ECOG 0 or 1
8. Patients must be willing to practice birth control from the time of enrollment on this study and for 12 months after the last dose of combined chemotherapy for women and for four months after treatment for men..
9. Women of child-bearing potential must be willing to undergo a pregnancy test prior to the start of treatment because of the potentially dangerous effects of the treatment on the fetus.

   NOTE: Certain malignancies may secrete hormones that produce false positive pregnancy tests. Serial blood testing (e.g. HCG measurements) and/ or ultrasound may be performed for clarification.
10. Serology

    -Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive may have decreased immune-competence and thus may be less responsive to the experimental

    treatment and more susceptible to its toxicities.)

    -Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative
11. Hematology

    * ANC > 1000/mm^3 without the support of filgrastim
    * WBC greater than or equal to 2500/mm^3
    * Platelet count greater than or equal to 80,000/mm^3
    * Hemoglobin > 8.0 g/dL. Subjects may be transfused to reach this cut-off.
12. Chemistry

    * Serum ALT/AST less than or equal to 5.0 x ULN
    * Serum creatinine less than or equal to 1.6 mg/dL
    * Total bilirubin less than or equal to 2.0 mg/dL, except in patients with Gilbert s Syndrome, who must have a total bilirubin < 3.0 mg/dL.
13. Patients must have completed any prior systemic therapy at the time of enrollment.

    Note: Patients may have undergone minor surgical procedures or limited field radiotherapy within the four weeks prior to enrollment, as long as related major organ toxicities have recovered to less than or equal to grade 1.
14. Ability of subject to understand and the willingness to sign a written informed consent document.
15. Willing to sign a durable power of attorney.
16. Subjects must be co-enrolled on the protocol 03C0277.

EXCLUSION CRITERIA:

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
2. Concurrent systemic steroid therapy.
3. Active systemic infections requiring anti-infective treatment, coagulation disorders, or any other active or uncompensated major medical illnesses.
4. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
5. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune-competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
6. History of severe immediate hypersensitivity reaction to cyclophosphamide, fludarabine, or aldesleukin.
7. History of coronary revascularization or ischemic symptoms.
8. For select patients with a clinical history prompting cardiac evaluation: last known LVEF less than or equal to 45%.

I. For select patients with a clinical history prompting pulmonary evaluation: known FEV1 less than or equal to 50%.

j. Patients who are receiving any other investigational agents.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-05-16 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Response rate | 6 weeks and 12 weeks following administration of the cell product, then every 3 months x3, then every 6 months x 2 years, then per PI discretion
  Percentage of patients who have a clinical response (PR+CR) to treatment (objective tumor regression)
Frequency and severity of treatment-related adverse events | From time of cell infusion to two weeks after cell infusion
  Grade and type of toxicity per dose level; fraction of patients who experience a DLT at a given dose level, and number and grade of each type of DLT

CONTACTS AND LOCATIONS:
Overall Officials: James C Yang, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Abrams SI, Khleif SN, Bergmann-Leitner ES, Kantor JA, Chung Y, Hamilton JM, Schlom J. Generation of stable CD4+ and CD8+ T cell lines from patients immunized with ras oncogene-derived peptides reflecting codon 12 mutations. Cell Immunol. 1997 Dec 15;182(2):137-51. doi: 10.1006/cimm.1997.1224. PMID 9514698
- [Background] Davis JL, Theoret MR, Zheng Z, Lamers CH, Rosenberg SA, Morgan RA. Development of human anti-murine T-cell receptor antibodies in both responding and nonresponding patients enrolled in TCR gene therapy trials. Clin Cancer Res. 2010 Dec 1;16(23):5852-61. doi: 10.1158/1078-0432.CCR-10-1280. PMID 21138872
- [Background] Wang QJ, Yu Z, Griffith K, Hanada K, Restifo NP, Yang JC. Identification of T-cell Receptors Targeting KRAS-Mutated Human Tumors. Cancer Immunol Res. 2016 Mar;4(3):204-14. doi: 10.1158/2326-6066.CIR-15-0188. Epub 2015 Dec 23. PMID 26701267
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-C-0017.html